CLINICAL TRIAL: NCT00384202
Title: A Multicenter, Open, Single Sequence Crossover Study to Assess the Safety and Efficacy of a Tacrolimus Modified Release, FK506E (MR4), Based Immunosuppressive Regimen in Stable Liver Transplant Patients Converted From a Prograf® Based Immunosuppressive Regimen
Brief Title: A Conversion Study to Assess Safety and Efficacy of a MR4 Based Immunosuppressive Regimen in Stable Liver Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMR-EC-1105
Record Dates: First submitted 2006-10-04; First posted 2006-10-05 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Transplantation
Keywords: Tacrolimus; Liver Transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Immunosuppression
  Other Names: Advagraf, FK506E, MR4

SUMMARY:
Assessment of the safety and the efficacy of a tacrolimus modified release (MR4) based immunosuppressive regimen in stable liver transplant subjects converted on a 1:1 (mg:mg) basis from a Prograf® based immunosuppressive regimen.

DETAILED DESCRIPTION:
Multicenter, open, single sequence crossover study. Subject Enrolment: Prograf® administered twice daily is replaced by Prograf as study medication, administered twice daily.

Six weeks Prograf-Treatment Phase to confirm compliance to regimen stability requirements (see Inclusion and Exclusion Criteria), and collection of data under Prograf treatment.

Conversion from Prograf (twice daily, morning & evening dosing) total daily dose to MR4 once daily (only morning dosing) on a 1:1 (mg:mg) basis on Day 1.

Twelve weeks MR4-Treatment Phase with study assessments for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant at least 12 months prior to enrollment.
* Prograf® dose remained unchanged for a minimum of 12 weeks prior to enrollment and tacrolimus whole blood trough level measurements were in the range of 5-15 ng/mL.

Exclusion Criteria:

* Any unstable medical condition that could interfere with the study objectives in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Creatinine clearance | 12 weeks

SECONDARY OUTCOMES:
Blood pressure, HbA1c, Acute rejection episodes | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma GmbH
Locations (13):
- France (3):
  - Lyon
  - Strasbourg
  - Villejuif
- Germany (2):
  - Berlin
  - Hamburg
- Dublin, Ireland
- Warsaw, Poland
- Spain (5):
  - Barakaldo
  - Barcelona
  - Santiago de Compostela
  - Seville
  - Valencia
- Birmingham, United Kingdom